CLINICAL TRIAL: NCT00673426
Title: Safety Evaluation of Use Sodic Enoxaparin Produced by the Laboratory Blausiegel When Compared With Product Clexane of Sanofi-Aventis Ltda in Chronic Renal Desease Patients.
Brief Title: Safety Evaluation of Use Sodic Enoxaparin
Acronym: Enoxaparin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ENOBLA0108
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-01

CONDITIONS: Kidney Disease
Keywords: enoxaparin; chronic renal disease; Anticoagulant activity of enoxaparin sodic
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Biological: Enoxaparin sodic

INTERVENTIONS:
Biological: Enoxaparin sodic

SUMMARY:
The purpose of this study was to evaluate safety, not inferiority clinical and pharmacodynamic profile of the drug Enoxaparin Sodium produced by laboratory Blausiegel when compared with Clexane product, produced by Laboratory Sanofi-Aventis in 60 patients with Chronic Renal Desease.

DETAILED DESCRIPTION:
Hemodialysis is a filtering and cleaning process of endogenous and exogenous metabolic blood products. The level control of anticoagulants in patients with chronic renal disease is indispensable. Evidence of clotting as TTPa and evidence of activity of anti-factor Xa should be used as a substrate to protect these patients, undergoing dialysis. The Enoxaparin sodium is one that acts as antithrombin-factor Xa inhibitor of acting directly on the inactivation of antithrombin. Thus, small-chain molecules (low molecular weight) as Enoxaparin show fundamentally anti-Xa high end and low end antitrombotic. The purpose of this study was to evaluate safety, not inferiority clinical and pharmacodynamic profile of the drug Enoxaparin Sodium produced by laboratory Blausiegel when compared with Clexane product, produced by Laboratory Sanofi-Aventis in 60 patients with Chronic Renal Desease. The study was kind of parallel, randomized, double-blind and systematic sampling. The drugs were administered during 12 consecutive dialysis sessions at a dose of 1 mg / kg. The activity of the drugs was verified by the strength of markers TTPa and anti-Xa and security was seen through adverse reactions and the evaluation function of capillaries.

The study was conducted 60 patients with chronic renal desease to both sexes, above 18 years aged, who were carrying out haemodialysis treatment during 3 times a week and satisfied inclusion criteria. The investigational products were randomly administered to patients in 12 consecutive dialysis sessions, at a dose of 1 mg / kg. The primary endpoint was safety of using the drug evaluated by monitoring events as:

* Loss of blood clotting by the system
* Blood coagulation and loss of capillary vein.
* Thrombus of capillary in 3 sessions of monitoring.
* Increase in the patient's hematocrit
* Thrombocytopenia
* Hematoma
* Fever
* Allergic reactions

The secondary endpoint was evaluation of non inferiority clinic, observed over the criteria in maintaining the non-coagulation of the extracorporeal circuit during hemodialysis and the pharmacodynamic curve effect of enoxaparin sodium verified by the strength of markers TTPa, anti-Xa and anti-IIa.

ELIGIBILITY:
Inclusion Criteria:

* Adults of both sexes, regardless of colour or social class;
* Above 18 years age, with good clinical features, to medical criterion;
* Patients who agreed to participate and signed the Informed Consent;
* Patients with Chronic Kidney Disease in hemodialysis treatment (3 times per week);
* Patients with clearance of creatinine <30ml/min;
* Patients with details of anticoagulants during hemodialysis.

Exclusion Criteria:

* Not agree to the terms described in Informed Consent;
* Volunteers bearers of the sensitivity enoxaparin sodium;
* Volunteers Patients with hypersensitivity to benzyl alcohol;
* Volunteers with a history of bleeding or disease that change of blood clotting could aggravate or terminate the clinical picture, such as tables of gastric ulcer;
* Volunteers with a history of peptic ulcer;
* Patients with body mass index greater than 30;
* Patients with cancer because of the possibility of compromising the function of the variable clotting;
* Patients in a period of post-pregnancy or childbirth;
* Patients with genetic abnormality of the system of coagulation;
* Polytraumatized patients;
* Patients in use of glucocorticoids for at least 1 month;
* Patients in use of other anticoagulants;
* Patients with high rate of bleeding;
* Patients undergo any surgery performed less than 15 days due to the risk of the formation of bruising at the site of surgery.
* Hypertension above 140/90 mmHg
* Patients in use of medicines could affect the hemostasis

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-01; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica TOP Nefrologia e Diálise, Americana, Brazil